CLINICAL TRIAL: NCT06675396
Title: Cohort Study on the Psychiatric Outcomes and Genetic Associations in Patients With Chronic Kidney Disease
Brief Title: Pharmacogenomics of Mood Disorder in Chronic Kidney Disease Patients
Acronym: CKD
Status: Not yet recruiting | Type: Observational
Sponsor: Wonju Severance Christian Hospital (Other)
Responsible Party: Principal Investigator, Jun Young Lee, Professor, Wonju Severance Christian Hospital
Other Study IDs: CKD gene; CKD Research Institute (Other: Wonju Severance Christian hospital)
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Chronic Kidney Disease(CKD); Depression
Keywords: CKD; Mood disorder
MeSH Terms: conditions — Renal Insufficiency, Chronic; Depression; Mood Disorders | interventions — Antidepressive Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Whole genome analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- chronic kidney with mood disorder: Patients developed mood disorder after chronic kidney disease development
  Interventions: Other: Antidepressants

INTERVENTIONS:
Other: Antidepressants — control

SUMMARY:
By using genetic information we could predict the prevalence of mood disorder and response to treatment.

DETAILED DESCRIPTION:
This prospective cohort study enrols patients with chronic kidney disease and gathers genetic information. By the patient's biochemical information, including genetic information, we could predict the prevalence of mood disorder and response to the antipsychotherapy.

ELIGIBILITY:
Inclusion Criteria:

* CKD patients aged 18 to 90 years

Exclusion Criteria:

* no CKD patients, aged below 18 or above 90 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CKD without history of mood disorder
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of depression | 10 years
  Prevalence of depression

IPD SHARING:
Plan to Share IPD: No